CLINICAL TRIAL: NCT00108225
Title: 2895 Effect of a High Protein Diet on the 24-hr Profile of Ghrelin, GH and IGF-1
Brief Title: Effect of a High Protein Diet on the 24-hour Profile of Ghrelin, GH (Growth Hormone) and IGF-1 (Insulin-like Growth Factor-1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03448-A
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Cholesterol; Creatinine Clearance; Diabetes; Glycohemoglobin; High Protein Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): 30% carbohydrate, 30% protein, 40% fat
  Interventions: Other: LoBag Diet - test phase
- Arm 2 (Placebo Comparator): 55% carbohydrate, 15% protein, 30% fat
  Interventions: Other: LoBAG Diet - control phase

INTERVENTIONS:
Other: LoBag Diet - test phase — A Low Biologically Available Glucose (LOBAG30), weight maintaining diet consisting of 30% carbohydrate, 30% protein, 40% fat will be provided to subjects for 5 weeks.
  Arms: Arm 1
Other: LoBAG Diet - control phase — A control, weight maintaining diet consisting of 55% carbohydrate, 15% protein, 30% fat will be provided to subjects for 5 weeks
  Arms: Arm 2

SUMMARY:
In this study we tested the hypothesis that an increase in protein content of the diet will result in an increase in the 24-hour integrated circulating growth hormone (GH) and insulin-like growth factor-1 (IGF-1) concentrations and an increase in lean body mass in people with untreated type 2 diabetes.

DETAILED DESCRIPTION:
Subjects with untreated type 2 diabetes were studied using a randomized crossover design. The study began with an initial two-week observation period. Subjects then were randomly assigned to one arm of the study for 5 weeks. The carbohydrate:protein:fat ratio for the control diet is 55:15:30 whereas for the test diet it is 40:30:30. Following a five-week washout period, subjects were assigned to the other arm of the study. All meals were provided by the SDTU. A six-day rotating meal plan has been devised. At the beginning and end of the 5-week diet period, the subject was admitted to the SDTU (Special Diagnostic and Treatment Unit), was provided with the meals appropriate for the test or control arm of the study, and had blood drawn at various times during a 24-hour period. In addition to measurement of GH and IGF-1, IGF-binding proteins 1 and 3, ghrelin, and body composition were determined.

ELIGIBILITY:
Inclusion Criteria:

* People ages 55 - 75 years old with type 2 diabetes, not receiving oral hypoglycemic agents or insulin.
* Fasting plasma glucose < 250 mg/dl (<14 mM) (tGHb < 14%).

Exclusion Criteria:

* Subjects will be screened for hematological abnormalities, liver disease, kidney disease, macroalbuminuria (>300 mg/24 hours), untreated thyroid disease, congestive heart failure, angina, life-threatening malignancies, proliferative retinopathy, diabetic neuropathy, peripheral vascular disease, serious psychological disorders, a body mass index > 35, and a fasting triglyceride of > 400 mg/dl.
* Presence of any of the above will be considered exclusion criteria.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
IGF-1, GH, Body Composition | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gannon, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Medical Center, Minneapolis, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Gannon MC, Nuttall FQ. Effect of a high-protein diet on ghrelin, growth hormone, and insulin-like growth factor-I and binding proteins 1 and 3 in subjects with type 2 diabetes mellitus. Metabolism. 2011 Sep;60(9):1300-11. doi: 10.1016/j.metabol.2011.01.016. Epub 2011 Mar 15. PMID 21406307
- [Result] Nuttall FQ, Gannon MC. Effect of a LoBAG30 diet on protein metabolism in men with type 2 diabetes. A Randomized Controlled Trial. Nutr Metab (Lond). 2012 May 20;9(1):43. doi: 10.1186/1743-7075-9-43. PMID 22607113